CLINICAL TRIAL: NCT01196819
Title: A Prospective Multi-center Randomized Trial Assessing the Safety and Effectiveness of Biodegradable Polymer Target Release Rapamycin-Eluting STent vs. XIENCE V Everolimus-Eluting Stent for the Treatment of Coronary Artery Disease
Brief Title: Randomized MicroPort's Firehawk DES Versus Xience V: TARGET I Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Target I
Record Dates: First submitted 2010-09-06; First posted 2010-09-08 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xience V (Active Comparator): Implantation of Xience V drug eluting stent
  Interventions: Device: Xience V
- Firehawk (Experimental): Implantation of Firehawk drug eluting stent
  Interventions: Device: Firehawk

INTERVENTIONS:
Device: Firehawk — Implantation of Firehawk drug eluting stent
  Arms: Firehawk
Device: Xience V — Implantation of Xience V drug eluting stent
  Arms: Xience V

SUMMARY:
The purpose of this study is to evaluate new generation drug eluting stent (DES) of MicroPort of its safety, efficacy and delivery system in treating CAD.

DETAILED DESCRIPTION:
The primary endpoint is in-stent late lumen loss after 9 months of the stent implantation. The secondary endpoint is in-stent percent diameter stenosis.This study is based on non-inferior assumption (vs. Xience V), requiring both endpoints reach statistical significance. Prespecified OCT follow-up is planned at 3-Year after index procedure at 3 chosen hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75, male or women who are not pregnant
* Evidence of non-symptomatic ischemia, stable or non-stable angina or past heart attack cases
* Target lesion is primary, single artery and single lesion of coronary artery
* Target lesion vessel length ≤24mm, diameter 2.25mm-4.0mm
* Lesion diameter stenosis ≥70%
* Candidates understand the study, willing to sign Consent of Agreement and to willing to accept follow-up For long lesion group, at least one target lesion length ≥28mm，diameter 2.5mm-4.0mm, and one lesion needs to implant 33mm 0r 38mm long stent

Exclusion Criteria:

* Acute heart attack within one week
* Chronic complete stenosis (TIMI 0), left main lesion, three branches need to treat, branch vessel diameter ≤2.5mm and bypass lesion
* Calcified lesion failed in pre-dilation and twisted lesion
* In-stent restenosis
* Stent implanted within one year
* Severe heart failure (NYHA above III) or left ventricle EF <40%
* Renal function damage, blood creatinine >2.0mg/dl
* Bleeding risk; allergic to drugs and agents used in procedure/treatment
* Life expectation < 12 months
* No compliances to the protocol
* Heart implantation cases

Pre-specified OCT inclusion/exclusion criteria:

* Patients underwent 9-month angio F/U
* No binary restenosis at 9-month
* LLL between -0.01~0.2mm
* No mix-implanted stent
* No more than one bail-out stent
* No TLR occurred at 3 years after PCI
* The target vessel able to deliver the OCT catheter

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Pro & MD, Principal Investigator — Fuwai Hospital, Beijing, China
Locations (1):
- Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li CJ, Xu B, Guan CD, Gao RL; TARGETⅠTrial Investigators. [Long term safety and efficacy of a novel abluminal groove-filled biodegradable polymer sirolimus-eluting stent for the treatment of coronary de novo lesions]. Zhonghua Xin Xue Guan Bing Za Zhi. 2017 Nov 24;45(11):940-947. doi: 10.3760/cma.j.issn.0253-3758.2017.11.009. Chinese. PMID 29166720
- [Derived] Gao Z, Zhang R, Xu B, Yang Y, Ma C, Li H, Chen S, Han Y, Yuan Z, Lansky AJ, Guan C, Leon MB, Gao R; TARGET Investigators. Safety and efficacy of a novel abluminal groove-filled biodegradable polymer sirolimus-eluting stent for the treatment of de novo coronary lesions: two-year results from a prospective patient-level pooled analysis of TARGET trials. Catheter Cardiovasc Interv. 2015 Mar;85 Suppl 1:734-43. doi: 10.1002/ccd.25861. Epub 2015 Feb 19. PMID 25678281
- [Derived] Gao RL, Xu B, Lansky AJ, Yang YJ, Ma CS, Han YL, Chen SL, Li H, Zhang RY, Fu GS, Yuan ZY, Jiang H, Huo Y, Li W, Zhang YJ, Leon MB; TARGET I Investigators. A randomised comparison of a novel abluminal groove-filled biodegradable polymer sirolimus-eluting stent with a durable polymer everolimus-eluting stent: clinical and angiographic follow-up of the TARGET I trial. EuroIntervention. 2013 May 20;9(1):75-83. doi: 10.4244/EIJV9I1A12. PMID 23685298

RESULTS

PARTICIPANT FLOW:
Groups:
- Xience V DES as Comparative Arm: Use Xience V DES as control group
  DES implantation: Implant DES for CAD cases
- MicroPort Firehawk DES: Use MicroPort's new generation of Firehawk drug eluting stent
  DES implantation: Implant DES for CAD cases
Period: Overall Study
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Started | 231 | 227
Completed | 225 | 227
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES | Total
Number analyzed (Participants) | 231 | 227 | 458
Age, Continuous [Median (Standard Deviation); unit: years] | 59.97 (9.39) | 58.95 (9.42) | 59 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 70 | 143
  Male | 158 | 157 | 315
Region of Enrollment [Number; unit: participants]
  China | 231 | 227 | 458

OUTCOME MEASURES:

1. Primary Outcome: 9 Months In-stent Late Lumen Loss
Description: To observe in-stent late lumen loss after 9 months of stent implantation It means the difference between the minimal lumen diameter immediately after stent implantation and the minimal lumen diameter by angiography review 9 months after the procedure
Time Frame: 9 months
Population: Angiographic follow-up at nine months was completed in 87.6% (199/227) of the Firehawk DES group and 87.4% (202/231) of the Xience V DES group.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Number analyzed (Participants) | 202 | 199
mm | 0.13 (0.18) | 0.13 (0.24)
Statistical Analysis 1: Comparison: Xience V DES as Comparative Arm vs MicroPort Firehawk DES; H0: Pe - Pc≥ ∆, H1: Pe - Pc < ∆. Pe and Pc are the mean 9-month in-stent late loss for the subject in the Firehawk DES group and the Xience group, respectively. ∆ is the non-inferiority margin. A two-sided upper 95% confidence bound will be calculated for the difference in 9-month in-stent late loss; Test type: Non-Inferiority — Non-inferiority margin is 0.13mm, if the two-sided upper 95% confidence bound is <Δ, the Firehawk Stent being tested will be considered non-inferior to the control. This corresponds to a P value <0.05 from a two-sided Student t-test comparing the difference between FirehawkStent and Xience stent to delta; p = 0.94, ANCOVA; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0 to 0.29]

2. Secondary Outcome: 9 Months In-stent Diameter Stenosis
Description: the in-stent diameter stenosis 9 months post-procedure
Time Frame: 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of diameter stenosis
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Number analyzed (Participants) | 202 | 199
percentage of diameter stenosis | 11.51 (7.37) | 11.85 (9.67)
Statistical Analysis 1: Comparison: Xience V DES as Comparative Arm vs MicroPort Firehawk DES; Test type: Non-Inferiority — Assume the in-stent percent diameter stenosis of both FIREHAWK and XIENCE V are 16 ± 16%, the non-inferiority value is 5%, the level of statistical significance is 0.05 (bilateral test), the power is 85%; p = 0.69, Mixed Models Analysis

3. Secondary Outcome: Target Lesion Failure(TLF) Rate
Description: Percentage of participants with the determination of TLF. TLF is the composite of sudden cardiac death, target vessel myocardial infarction, and ischemic driven target lesion revascularization (TLR).
Time Frame: 1 years after index PCI
Measure: Number; unit: percentage
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Number analyzed (Participants) | 231 | 227
percentage | 2.2 | 2.2
Statistical Analysis 1: Comparison: Xience V DES as Comparative Arm vs MicroPort Firehawk DES; Test type: Other; p = 1.0, Fisher Exact

4. Secondary Outcome: TLF(Target Lumen Failure) Rate
Description: percentage of participants with the determination of TLF, TLF include target vessel myocardial infarction, symptom-driven target lesion revascularization and sudden cardiac death.
Time Frame: 3 years after index PCI (Percutaneous Coronary Intervention)
Population: 3 patients in Xience V DES group and 5 patients in Firehawk DES group failed to be contacted.
Measure: Number; unit: percentage
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Number analyzed (Participants) | 228 | 222
percentage | 3.51 | 4.05
Statistical Analysis 1: Comparison: Xience V DES as Comparative Arm vs MicroPort Firehawk DES; Test type: Other; p = 0.76, Fisher Exact

5. Secondary Outcome: TLF(Target Lumen Failure)
Description: as for outcome 4
Time Frame: 5 years after index PCI
Population: 6 patients in Xience V DES group and 10 patients in Firehawk DES group failed to be contacted.
Measure: Number; unit: percentage
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Number analyzed (Participants) | 225 | 217
percentage | 6.67 | 5.99
Statistical Analysis 1: Comparison: Xience V DES as Comparative Arm vs MicroPort Firehawk DES; Test type: Other; p = 0.77, Fisher Exact

6. Secondary Outcome: Number of Participants With Stent Thrombsis (ARC Defined Definite/Probable)
Time Frame: 1 years after index PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Number analyzed (Participants) | 231 | 227
Participants | 0 | 0
Statistical Analysis 1: Comparison: Xience V DES as Comparative Arm vs MicroPort Firehawk DES; Test type: Other; p = 1.0, Fisher Exact

7. Secondary Outcome: Number of Participants With Stent Thrombsis (ARC Defined Definite/Probable)
Time Frame: 3 years after index PCI
Population: 3 patients in Xience V DES group and 5 patients in Firehawk DES group failed to be contacted.
Measure: Count of Participants; unit: Participants
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Number analyzed (Participants) | 228 | 222
Participants | 1 | 0

8. Secondary Outcome: Number of Participants With Stent Thrombsis (ARC Defined Definite/Probable)
Time Frame: 5 years after index PCI
Population: 6 patients in Xience V DES group and 10 patients in Firehawk DES group failed to be contacted.
Measure: Count of Participants; unit: Participants
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
Number analyzed (Participants) | 225 | 217
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Xience V DES as Comparative Arm | MicroPort Firehawk DES
All-Cause Mortality (participants affected / at risk) | 8/225 | 7/227
Serious Adverse Events (participants affected / at risk) | 46/225 | 28/227
Other Adverse Events (participants affected / at risk) | 0/225 | 0/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xience V DES as Comparative Arm (N=225) | MicroPort Firehawk DES (N=227)
death (Injury, poisoning and procedural complications) | 8 | 7
myocardial infarction (Cardiac disorders) | 9 | 5
coronary revascularization (Surgical and medical procedures) | 28 | 16
Definite/probable in-stent thrombosis (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No